CLINICAL TRIAL: NCT07108231
Title: Effects of Inspiratory Muscle Training on Inspiratory Muscle Strength in Hospitalized Heart Failure Patients: A Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training in Hospitalized Heart Failure Patients
Acronym: IMTHHF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CAROLINA NIGRO DI LEONE (Other)
Responsible Party: Sponsor-Investigator, CAROLINA NIGRO DI LEONE, Lead Physiotherapist, Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CAAE:88229525.1.0000.5259
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Inspiratory Capacity; Inspiratory Muscle Strength; Hospitalizations
Keywords: HEART FAILURE; EXERCISE INTOLERANCE; INSPIRATORY MUSCLE TRAINNING; HOSPITALIZATION
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a phase 1 randomized, controlled clinical trial with two arms.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): IMT group
  Interventions: Device: Inspiratory muscle trainning
- control (Sham Comparator): Sham
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Inspiratory muscle trainning — The IMT protocol will involve the use of the Power Breath® linear resistor device, classic light model (Anvisa Registration: 81001390001). The IMT group will perform the protocol with a load ranging from 30% to 50% of maximal inspiratory pressure (MIP). Two daily sessions of 30 repetitions each will be conducted, starting with a minimum load of 30%, with a 10-minute interval between sessions, and a proposed weekly load increase based on patient tolerance.
  For training load progression, patient effort will be taken into account, aiming to maintain a perceived exertion level between light and moderate fatigue (BORG scale less than 4).
  Patients will remain seated at a 90° angle, using a nasal clip, and will be encouraged to perform consecutive inspirations with their mouth on the device's mouthpiece. Vital signs-including blood pressure (BP), mean arterial pressure (MAP), peripheral oxygen saturation (SpO2), respiratory rate (RR), heart rate (HR)-and dyspnea sensat
  Arms: INTERVENTION
Device: Sham (No Treatment) — The control group (IMTsham) will perform two daily sessions of 30 repetitions each without any load, using the same resistor device.
  Arms: control

SUMMARY:
Introduction Exercise intolerance is the most common symptom in patients with heart failure (HF), significantly impacting their quality of life and functional capacity. Muscle metabolism may be impaired due to sympathetic hyperactivation, systemic inflammation, and neurohormonal alterations, contributing to ventilatory inefficiency and exercise intolerance. Inspiratory muscle training (IMT) has been shown to improve inspiratory muscle strength and endurance, reducing fatigue and the sensation of dyspnea.

There is a gap in the evidence regarding the use of IMT in hospitalized settings, particularly concerning short-term gains in inspiratory muscle strength and the safety of the intervention. This study aims to evaluate the effects of IMT on inspiratory muscle strength, hemodynamic and functional outcomes, as well as the safety of the IMT protocol in hospitalized patients with HF.

Methods A randomized, controlled clinical trial will be conducted in the Cardiac Intensive Care Unit of the University Hospital Pedro Ernesto. The study will include individuals of both sexes, aged 18 years or older, who are hospitalized due to heart failure.

Exclusion criteria will include: pregnancy; head trauma and/or brain injury; motor disability; signs and/or symptoms of low cardiac output; acute coronary syndrome; advanced HF with left ventricular ejection fraction (LVEF) below 20%; presence of untreated tachyarrhythmias or bradyarrhythmias; use of high-dose inotropes or vasopressors or an increase in their dose within the past 24 hours.

Primary outcomes will include inspiratory muscle strength, safety, functional status, length of stay in the ICU, and hospital readmission within 90 days. After randomization, the intervention group will undergo IMT with a load between 30% and 50% of maximal inspiratory pressure (MIP), while the control group will perform IMT without load.

It is expected that IMT will be safe and lead to improvements in inspiratory muscle strength and functional status, without significant hemodynamic repercussions.

DETAILED DESCRIPTION:
In hospitalized patients, the use of inspiratory muscle training (IMT) may be particularly beneficial to mitigate muscle strength loss caused by hospitalization, reduce length of stay, and optimize the transition to post-discharge rehabilitation. Thus, the implementation of IMT in the hospital setting can be a safe intervention capable of improving the functional capacity of patients with heart failure.

Despite the known benefits, to date there are no studies conducted with heart failure patients admitted to intensive care units that evaluate gains in inspiratory muscle strength and their hemodynamic and functional effects.

After recruitment, patients will be randomized (using the website random.org) into an Intervention group, which will perform inspiratory muscle training (IMT), and a Control group, which will perform a sham IMT (IMTsham). Both groups will follow the institutional ICU rehabilitation protocol.

The IMT protocol will involve the use of the Power Breath® linear resistor device, classic light model (Anvisa Registration: 81001390001). The IMT group will perform the protocol with a load between 30% and 50% of maximal inspiratory pressure (MIP). Two daily sessions of 30 repetitions each will be conducted, starting with a minimum load of 30%, with a 10-minute interval between sessions, and with a proposed weekly load increase according to patient tolerance.

For training load progression, patient effort will be considered, aiming to maintain a perceived exertion level between light and moderate fatigue (BORG scale less than 4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure;
* age over 18 years;
* hospital admission due to heart failure;
* clinical and hemodynamic stability defined as: heart rate > 40 bpm and < 130 bpm; systolic blood pressure (SBP) > 90 mmHg and < 180 mmHg; mean arterial pressure (MAP) > 60 mmHg and < 110 mmHg; respiratory rate > 5 breaths per minute and < 40 breaths per minute; peripheral oxygen saturation > 88%; absence of psychomotor agitation or somnolence

Exclusion Criteria:

* pregnancy;
* head trauma and/or brain injury;
* motor incapacity preventing participation in the institutional rehabilitation protocol of the Cardiointensive Care Unit (ICU);
* signs and/or symptoms of low cardiac output (such as sweating, hypotension, hyperlactatemia, nausea);
* acute coronary syndrome;
* advanced heart failure with left ventricular ejection fraction (LVEF) less than 20%
* presence of untreated tachyarrhythmias or bradyarrhythmias;
* use of inotropes or vasopressors at high doses or dose escalation in the last 24 hours (dobutamine above 15 mcg/kg/min, milrinone above 0.5 mcg/kg/min, norepinephrine above 0.3 mcg/kg/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
inspiratory muscle strenght | Day 1, after 7 days of admission, through study completion, an average of 10 days
  Inspiratory muscle strength refers to the force generated by the muscles involved in inhalation, primarily the diaphragm and accessory respiratory muscles. It reflects the ability of these muscles to overcome resistance and expand the lungs during breathing. Before the tests to assess static and dynamic inspiratory muscle strength, volunteers underwent a familiarization session with the devices and maneuvers to be performed. After measuring resting hemodynamic parameters, the evaluation of maximal static respiratory pressures was conducted. Maximal inspiratory pressure (MIP) was measured using an analog manovacuometer (MURENAS brand, Anvisa Registration: 80244900005), following the protocol of the American Thoracic Society and the European Respiratory Society.
  MIP was determined after a maximal inspiratory effort starting from residual volume against airway occlusion.

SECONDARY OUTCOMES:
Assessment of Functional Status | Admission day, through study completion, an average of 10 days
  For the assessment of functional status, the 1-minute sit-to-stand test (1MSTS) will be performed. Participants will be instructed to stand up and sit down as quickly as possible without using their arms for 1 minute and will be advised to stop whenever they wish, if necessary. Heart rate (HR), respiratory rate (RR), blood pressure (BP), peripheral oxygen saturation (SpO2), and assessments of dyspnea and leg fatigue using the Modified Borg Scale will be recorded before and after the test. One repetition is defined as standing up fully straight and returning to a seated position.
Peripheral Muscle Strength | Admission day and through study completion, an average of 10 days
  Peripheral muscle strength (PMS) will be measured using a digital dynamometer (Digital Dynamometer MG4800). Volunteers will perform the maneuver seated at a 90-degree angle, with the elbow flexed at 90 degrees and the wrist in a neutral position. They will be instructed and encouraged to perform a maximal handgrip contraction for 3 seconds on both sides. Three maximal isometric contractions will be performed, and the highest value from the dominant hand will be used for analysis . Predicted normal values will be based on the reference equation for dominant upper limb grip strength in middle-aged and elderly Brazilians. Values below 70% of the predicted will be considered reduced peripheral muscle strength .
Adverse events | Through study completion, an average of 10 days
  The safety of the IMT protocol will be evaluated by monitoring the occurrence of any adverse events during the intervention. Adverse events will be classified as mild, moderate, or severe (Table 1). The control group will also have adverse events recorded. The heterogeneity in the definition of safety criteria and adverse events is a limitation in the literature, due to the lack of standardization in the definitions and naming of adverse events in clinical practice . Mild events are considered transient and do not require clinical intervention. Moderate events cause temporary symptoms that require clinical intervention. Severe events are those that result in permanent sequelae, serious complications, or even life-threatening conditions, such as cardiac arrest, loss of consciousness, and death .During the intervention period, hemodynamic effects of IMT will be assessed by monitoring vital signs before and after protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Nigro Di Leone, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes